CLINICAL TRIAL: NCT01175551
Title: Direct Measurements of Cervical Remodeling for Predicting Preterm Birth
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Burroughs Wellcome (Industry); Bayer Droegemueller Award in Clinical Research (Unknown)
Responsible Party: Principal Investigator, Michal A. Elovitz, Associate Professor, Director, Maternal and Child Health Research Program, Department of Obstetrics and Gynecology, University of Pennsylvania
Other Study IDs: 810707
Record Dates: First submitted 2010-07-29; First posted 2010-08-05 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Preterm Birth
Keywords: Preterm Birth; Cervix; Cervical Shortening; Cervical remodeling; PTB
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — maternal serum, maternal cervical vaginal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: women screened at Penn OB/GYN Associates or Helen O. Dickens Center with a documented singleton pregnancy less than 18 weeks gestational age
- Group 2: Nulliparous pregnant women (no previous pregnancy greater than 15 weeks) screened at Penn OB/GYN Associates or Helen O. Dickens Center less than 18 weeks gestational age

SUMMARY:
Racism and health care system distrust are potent stressors and may be associated with preterm birth (PTB). Additionally, cervical shortening is a common pathway leading to PTB. This study is enrolling a prospective cohort of pregnant women. The study assesses racial discrimination, health care system distrust, and cervical change using 2 questionnaires, exam, and protein levels in cervical vaginal fluid and maternal serum.

DETAILED DESCRIPTION:
Preterm birth (PTB) is currently the most important maternal and child health problem in the United States. It is the leading cause of neonatal mortality and a significant contributor to neonatal morbidity. In the United States, approximately 12% of all live births are born preterm, an incidence that continues to rise. The extreme cost of PTB resides not only in the immediate neonatal care but also in the longterm care of lasting morbidities resulting from prematurity. Effective prevention or treatment of PTB could significantly lower neonatal mortality and morbidity as well as health care costs. In the United States, PTB costs on the order of 28 billion dollars a year. But, this cost does not stop at the delivery. The costs of prolonged hospital care after birth and the increased need for hospital admission during the first year of life for ex-preterm infants is significant and confers a large economic burden on our society.

It is well known that PTB rates in the United States are highest for Black infants (17.9%), followed by Native Americans (14%), White infants (11.8%), and Asian infants (10%). The specific large disparity between black and white infants is striking and the etiology of this disparity is not fully understood. This disparity persists even after adjusting for socioeconomic status. Maternal stress has been implicated as a potential cause of PTB. Racism is a potent lifetime stressor in the lives of Black women in particular. It is plausible that perceptions of racism as well as distrust in the health care system may explain the persistent racial disparities in PTB, especially through mediation of other factors associated with premature birth. The data to date offer a preventative strategy only to those women with a prior PTB. These women represent a small percent of all women with a PTB. More then half of all PTB occur in apparently low risk pregnancies. Cervical shortening appears to be a common biological pathway leading to preterm birth, often well in advance of PTB. Regardless of etiology of PTB, cervical change must occur. The cervix must remodel (change) for birth to occur at any gestational age.

We hypothesize that experiences of discrimination and health care system distrust are associated with preterm birth. Further, we hypothesize that premature cervical remodeling occurs weeks prior to actual birth and may be able to be detected in women at highest risk for preterm birth (nulliparous women-women who have not previously carried a pregnancy beyond 15 weeks). This study investigates whether experiences of discrimination and health care system distrust are associated with PTB in all women (group 1). It also investigates if the detection of cervical remodeling (changes in the cervix measured by protein levels, ultrasound length and physical exam) can accurately identify those women at greatest risk for PTB-nulliparous (group 2). A prospective cohort of pregnant women will be enrolled. All enrolled women are asked to complete validated questionnaires about experiences of discrimination and health care system distrust. Nulliparous women are evaluated for cervical change, through a comprehensive evaluation at 18-24 weeks. The main outcome assessed is preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women screened at < 18 weeks with a documented singleton pregnancy, who agree to participate in the study (group 1). A subset of Nulliparous women (no previous pregnancy 15 weeks)(group 2) will be assessed.
* Women of all races and age will be included.

Exclusion Criteria:

* Women with a multi-fetal pregnancy, current use of systemic steroids or immunosuppressive therapy or enrollment for prenatal care after 24 weeks.
* Women with a prior documented history of Leep or Conization will be excluded.
* Any known Mullerian anomalies such as septate uterus, bicornuate or unicornuate uterus will be excluded given that these are high risk groups for preterm delivery.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All pregnant women screened at Penn OB/GYN Associates or Helen O. Dickens Center at less than 18 weeks gestational age with a documented singleton pregnancy who agree to participate in the study (group 1); Nulliparous women (no previous pregnancy greater than 15 weeks)less than 18 weeks gestational age (group 2)
Sampling Method: Non-Probability Sample
Enrollment: 1207 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Preterm birth (delivery at less than 37 weeks) | up to 42 weeks
  16-37 weeks from enrollment

SECONDARY OUTCOMES:
spontaneous Preterm Birth at less than 37 weeks and less than 34 weeks, small for gestational age (less than the 10% birth weight for gestational age as determined by the Alexander curve), preeclampsia and a composite of neonatal outcomes | up to 42 weeks
  16-37 weeks from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Michal A Elovitz, MD, Principal Investigator — University of Pennsylvania; Sindhu Srinivas, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Helen O. Dickens Center for Women, Philadelphia, Pennsylvania
  - Penn OB/GYN Associates, Philadelphia, Pennsylvania